CLINICAL TRIAL: NCT02912962
Title: Self-Regulation in Adolescents With FASD: The Efficacy of a Targeted Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Glenrose Foundation (Other); Woman and Children's Health Research Institute (Unknown); NeuroDevNet (Other); Provincial Health Services Authority British Columbia (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00064830
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2017-10

CONDITIONS: Self-regulation; Adolescents; Fetal Alcohol Spectrum Disorder
MeSH Terms: conditions — Self-Control; Fetal Alcohol Spectrum Disorders

ARMS (2):
- Intervention Group (Experimental): Cognitive testing 1, 12 intervention sessions, Cognitive testing 2, Approximately a 12 week wait (no intervention), Cognitive testing 3.
  The intervention is a 12 week, individualized, one-on-one self-regulation intervention where adolescents will learn to attain, change, or maintain an appropriate level of alertness .
  Interventions: Behavioral: Self-Regulation Intervention adapted from the Alert Program ®
- Waitlist (Experimental): Cognitive testing 1, Approximately a 12 week wait (no intervention), Cognitive testing 2, 12 intervention sessions, Cognitive testing 3
  Interventions: Behavioral: Self-Regulation Intervention adapted from the Alert Program ®

INTERVENTIONS:
Behavioral: Self-Regulation Intervention adapted from the Alert Program ®

SUMMARY:
Fetal alcohol spectrum disorder (FASD) describes a collection of physical, mental, and behavioral disabilities that result from prenatal alcohol exposure (PAE). Individuals with FASD often struggle with self-regulation, or the ability to control thoughts, emotions and actions, which can lead to many long-term problematic life circumstances.

This study aims to improve self-regulation abilities in adolescents, aged 11-17, with FASD using a targeted intervention. Researchers adapted the Alert Program®, a developed intervention targeting self-regulation in children, to be appropriate for an adolescent FASD population. Participants are split into two groups: an FASD intervention group, and an FASD waitlist group. These groups are compared on a variety of measures. These measures include cognitive measures (executive functioning, response conflict, inhibitory control, etc), behavioural measures (self-regulation, adaptive behaviour, etc), and physiological measures (cortisol and sleep). The FASD intervention group will be tested at baseline and once after the intervention, and lastly after an approximately 12-week wait following the intervention. The FASD waitlist group will be tested at baseline, after a three month wait period, and again after receiving the intervention.

The investigators expect that the Alert program® will lead to significant improvements in participant's self-regulation abilities as evidenced by cognitive, behavioural, and physiological changes. Improving self-regulation in adolescents with FASD will reduce the high level of adverse outcomes experienced by adolescents with FASD, and help them have a successful transition into adulthood.

DETAILED DESCRIPTION:
Objectives:

The goal of the proposed research is to determine if adolescents with Fetal Alcohol Spectrum Disorder (FASD) will have improvements in their ability to self-regulate after the implementation of a targeted intervention. The project is part of the larger NeuroDevNet renewal grant. The goals of the proposed project are to study adolescents with FASD to examine: 1) the association of measures of Executive Function (EF) and self-regulation with life adversities and adverse outcomes 2) cortisol regulation in FASD and its association with life adversity and difficulties with EF, self-regulation, sleep, and adverse outcomes 3) whether EF, self-regulation, sleep, and cortisol regulation can be improved with an intervention targeting self-regulation.

Research questions:

Can self-regulation among adolescents with FASD be improved with a targeted intervention? The investigators hypothesize that the participants with FASD in the modified Alert Program ® intervention will have greater improvements on cognitive, behavioral, and physiological measures of self-regulation compared to the wait-list control group.

1. How is self-regulation impacted in adolescents with FASD? The investigators hypothesize that adolescents with FASD will have significantly lower scores (at baseline) on a variety of measures of self-regulation including cognitive, behavioral, and physiological measures (cortisol regulation and sleep behaviors) compared to normative samples. This information is important for informing the profile of self-regulation impairments in FASD.
2. Do improvements in self-regulation lead to improvements in functional outcomes of adolescents with FASD? The investigators hypothesize that following the intervention, participants with FASD will show improvements in reported functional outcomes on a measures adaptive functioning.

Background:

Individuals with FASD display significant executive functioning (EF) impairments (e.g., inhibition, decision making, thinking flexibly) as well as difficulties in regulating their behavior. They are at risk for early life adversities (e.g., unstable home environment) and adverse outcomes including mental health issues, delinquency, and substance abuse. Adverse outcomes in FASD may result from EF and self-regulation impairments that have the potential to be mitigated with targeted interventions. Altered hypothalamic-pituitary-adrenal (HPA) activity, as indexed by plasma cortisol levels, is a physiological marker of self-regulation. Importantly, PAE is known to affect HPA activity and regulation. Sleep behaviors are also disrupted in FASD, which is another physiological marker of self-regulation.

Recognizing the profile of self-regulation deficits in FASD, and the functional outcomes of such impairments will equip the investigators to examine the impact of intervention efforts on self-regulation. Research on the efficacy of interventions to improve various indices of self-regulation in FASD is critical, as this may then prevent later adverse outcomes. The Alert Program® is an evidence-based intervention program that focuses on self-regulation. It is a widely-used program that demonstrated some efficacy in children with FASD with improvements on parental reports of EF, behavioural and emotional regulation, and tests of social cognition, inhibitory control and emotional problem-solving. The investigators anticipate that this intervention, which has not been studied in adolescents with FASD, will lead to improvements across a range of self-regulatory functions including cognitive, behavioral, and physiological indicators.

Method:

Participants. FASD Group: Recruitment and data collection in Alberta will occur in Dr. Rasmussen's and Pei's research lab at the Glenrose Rehabilitation Hospital (GRH) and with Dr. Oberlander in the Child and Family Research Institute at the University of British Columbia (under a separate University of British Columbia ethics application). The GRH facility consists of testing rooms, offices, and workstations. Participants who have participated in previous research studies by Drs. Pei and Rasmussen will be informed about the study by a research assistant and will be provided an information letter. Parents will then have the opportunity to discuss the study further and set up an appointment with the research assistant or they may contact the lab at a later time should they choose to participate. Eligible participants not currently involve in the investigators' studies will receive an information letter from the FASD Clinic at the GRH describing the study to all eligible participants (in the mail or when they are seen by the clinic), who will be blinded from researchers. Interested caregivers will then contact the researchers if they want to participate, and the project coordinator will book testing sessions. For all cognitive assessments, a trained Research Assistant will administer assessment measures with participants while the caregiver completes questionnaires and rating scales. For those interested participants who have recently been involved in another study, cognitive test results will be shared between studies to minimize the baseline testing time for the participants, and reduce practice effects as some measures cannot be re-administered within a short time frame. Caregivers will also complete a 45-minute training module and worksheet (~15 minutes) at baseline testing. This training module will provide an overview of the program as well as discuss the five categories (mouth, move, touch, look and listen) that will form the base of the intervention strategies for their teen. An RA trained in the intervention who has access to Occupational Therapy consult will be conducting the interventions.

Procedure:

Study Design: All participants with FASD will be tested on the assessment battery at Baseline (Time 0) which will provide important information on the profile of self-regulation impairments in FASD, as well as baseline data against which efficacy of the intervention can be evaluated. The FASD group will then be divided into the targeted intervention group (Group A) and a waitlist control group (Group B) and both groups will be tested on the battery of tests after the intervention. The waitlist group will be tested once more after a waiting period, but before they receive the intervention. This mixed design allows the investigators to control for change due to development, practice effects, regression to the mean, and familiarity with the procedures. Rolling recruitment is required so that interventions are not all running at the same time, ensuring sufficient staff and resources to administer the interventions. The investigators feel it is important to provide the intervention to all participants using a waitlist design in a timely manner for ethical and clinical reasons.

The Alert Program® will be administered individually to participants by a trained RA or occupational therapist (e.g. post-doctoral fellow or a graduate student in Psychology or Occupational Therapy) in the investigators' lab space. A different RA will conduct all post intervention testing. Baseline testing will be conducted by the interventionist RA in order to establish a rapport and gain clinical knowledge to plan and individualize sessions to meet participants needs. The intervention is based on a teen adaptation of the Alert Program developed by Therapy Works Inc modified by the research team to meet the needs of adolescents with FASD. The intervention will consist of 12 one hour sessions that take place over the course of 9-15 weeks. Over the course of the 12 sessions the participants will work on moving through 3 stages (stage 1 - identifying engine speeds, stage 2- learning strategies to change engine levels, stage 3 - regulating engine speeds).

Measures: The investigators will be using a number of different measures for pre and post analysis of behavioural, cognitive, and physiological changes. The behavioural measures are: background questionnaire, Behavioural Rating Inventory of Executive Function (BRIEF)- 2, Monetary Choice Questionnaire, Dot-Probe Test of Attention Bias to Threat, Adolescent Self-Regulatory Inventory (ASRI), Adaptive Behaviour Rating System (ABAS)-2, Child Behavior Checklist (CBCL) (youth self-report, caregiver report), and The Stressful Urban Life Events Scale. The cognitive measures are: Wide Range Intelligence Test (WRIT), Delis-Kaplan Executive Function System (D-KEFS), Iowa Gambling Test (IGT), Whack-A-Mole Test, and the Rey Complex Figure Test. The physiological measures include both salivary cortisol and fingernail cortisol samples, and the Pediatric Sleep Questionnaire (PSQ).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study are adolescents ages 11-17 with confirmed prenatal alcohol exposure and an FASD diagnosis.
* The study includes participants with an Intelligence Quotient < 70 to allow for a range of cognitive abilities.

Exclusion Criteria:

* Exclusion criteria will include those with known genetic disorders (e.g., Down's syndrome), other severe neurodevelopmental disorders (e.g., autism) and significant motor/sensory impairments.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Delis-Kaplan Executive Function System (D-KEFS) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  a widely-used, normed measure of EF. Participants will complete the 2 subtests: trail making (cognitive flexibility and switching) and color-word interference (inhibition and switching).
Iowa Gambling Test (IGT) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  a computerized measure of decision making which involves behavioral and emotional regulation. Participants start with $2000 of theoretical money and have to choose cards one at a time from four decks (A, B, C, and D) to earn as much money as they can. There are two disadvantageous decks (large initial rewards and large losses) and two advantageous decks (small immediate rewards and smaller losses).
Whack-A-Mole Test | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  A computerized Go/NoGo paradigm will be used to measure inhibitory control, modeled after the "whack-a-mole" arcade game. Participants press a button every time a mole appears in monitored 'garden hole', but withhold responding when a garden vegetable appears. This task has been sensitive to interventions in previous studies of children with FASD.
Monetary Choice Questionnaire | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  Is a measure of affective decision making in children and a measure of hot EF. In this task participants will be asked to choose if they would rather a smaller amount of money now, or a larger amount later. Participants will be informed to answer as if they are actually receiving the money, but will be informed that the test is hypothetical, and they will not actually be receiving money on this task. This task is a form of measuring delay of gratification, where participants have to choose between a smaller award given immediately, or waiting and receiving a larger award. Performance on Delay of Gratification tests in early childhood is associated with academic, social, and mental well-being later on in life.
Dot Probe Task | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  Dot-probe task is a spatially oriented attention task that is administered via computer. The task aims to capture attentional bias toward emotional cues, and is primarily used to investigate threat-related attentional bias. Participants are briefly shown two stimuli, one threat-related and one neutral. They are then shown a small probe in the same location as one of the stimuli. Participants are required to respond as quickly as possible to the probe. Response times are thought to indicate the distribution of the participants' attention, with faster response times to probes in the attended to location. Attentional bias towards threat is demonstrated when participants attend quicker to probes that replace threat-related stimuli.
Rey Complex Figure Test (RCFT) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  The RCFT is a neuropsychological assessment tool that requires examinees to copy a complex geometric design with multiple embedded details, and then re-create the figure from memory. The tool places demands on many cognitive functions, including planning/organization, attention, visual-spatial perception and construction, motor ability, and memory encoding, storage, and retrieval processes. Evaluations of reliability and validity for the RCFT have proved excellent, with a median inter-rater reliability of .94. Based on the factor analyses, the RCFT appears to capture five domains of cognitive functioning: visuospatial recall memory, visuospatial recognition memory, response bias, processing speed, and visuospatial constructional ability.
Behavioral Rating Inventory of Executive Function- 2 (BRIEF-2) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  Caregivers will complete the BRIEF-2, a widely-used normed measure of EF including inhibition, set shifting, emotional control, working memory, planning, organization, and monitoring skills.
Adolescent Self-Regulatory Inventory (ASRI) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  The ASRI is self-report a measure of self-regulation (e.g. managing negative emotions, defer gratification) in adolescents.
Adaptive Behavior Assessment System (ABAS-2) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  The ABAS-II provides a comprehensive, norm-referenced assessment of the adaptive behavior and skills of individuals from birth to age 89.
Child Behavior Checklist (CBCL) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  The CBCL is a 117-item questionnaire that measures the competence and problem areas of children ages 6-18, as reported by caregivers and youth 11-18 years. The test yields scores in eight problem scales of behavioral and emotional problems labeled as: Withdrawn, Anxious/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Delinquent Behavior, and Aggressive Behavior. These scales can be summarized into three broader scales: Externalizing problems (Aggressive Behavior, Delinquent Behavior), Internalizing problems (Withdrawn, Somatic Complaints, Anxious/Depressed) and Total Problems. Scores are also given in three competence areas: social settings, activities, and school settings.
Health Habits Questionnaire | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  A 22 item self-report questionnaire focusing on the adolescent's preferences for physical activity, leisure, hobbies and interests, and sleeping habits (attached to ethics application). The information gathered from this questionnaire will be used to further individualize the intervention for the participant and will provide the interventionist with important information to assist in the improvement of self-regulation.
Paediatric Sleep Questionnaire (PSQ) | change from pre and post intervention (12 weeks), plus 3 month wait (waitlist group), and 3 month follow up (intervention group)
  The PSQ is a pen-and-paper parent questionnaire designed to screen for common sleep problems in children. The questionnaire includes 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric features.
Cortisol | Between Pre and Post intervention (12 weeks) 1) immediately upon awakening (AM sample); 2) within 30-minutes of bedtime (PM sample). Both salivary samples will be taken on two different days within a five-day period
  Two key indicators of HPA activity will be collected as physiological measures of self-regulation - the cortisol awakening response (CAR), and overall cortisol diurnal rhythm. Both cortisol diurnal rhythm and the CAR will be sampled at home.
Fingernail Cortisol | approximately 2-3 months
  The human stress response is regulated in part by the hypothalamic-pituitary-adrenal (HPA) axis. Activation of the HPA axis results in the release of cortisol and related steroids from the adrenal cortex. There are well-established techniques for measuring levels of cortisol using saliva, urine and blood. However, nail clipping is more acceptable under most circumstances, and nails are known for their resistance to decomposition and disintegration. A recent pilot study (Warnock et al., 2010) indicates that fingernail analysis allows one to assess accumulated hormone levels over a period of approximately 2-3 months, and thus analysis of fingernail cortisol could provide a novel measure of long-term HPA regulation/dysregulation in subjects in our proposed study.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia